CLINICAL TRIAL: NCT05239546
Title: Phase II, Single Arm Study of Neoadjuvant Dostarlimab (TSR-042) in Stage II and III Deficient Mismatch Repair Colon Cancers
Brief Title: Single Arm Study of Neoadjuvant Dostarlimab in Stage II and III Deficient Mismatch Repair Colon Cancers
Acronym: NAIO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Saima Sharif, Clinical Associate Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202105539
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Colon Cancer; dMMR Colorectal Cancer
Keywords: Colon cancer; dMMR; Deficient mismatch repair colon cancer; MSI-High; MSI-H; Non-operative management; No surgery
MeSH Terms: conditions — Colonic Neoplasms | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Dostarlimab (Experimental): Participants will receive Dostarlimab 500 mg IV every 3 weeks for 6 cycles followed by 1000 mg every 6 weeks for 8 cycles until 1.5 years
  Interventions: Drug: Dostarlimab

INTERVENTIONS:
Drug: Dostarlimab — Participants will receive Dostarlimab 500 mg IV every 3 weeks for 6 cycles followed by 1000 mg every 6 weeks for 8 cycles until 1.5 years
  Other Names: TSR-042

SUMMARY:
This is a Phase II, single arm study looking at the rate of major clinical response and non-operative management in Stage II and III colon cancer after 18 weeks (up to 6 cycles) of neoadjuvant dostarlimab.

DETAILED DESCRIPTION:
The purpose of this research study is to look at the effects of the immunotherapy drug dostarlimab on dMMR colon cancer tumors and to see if these patients can avoid surgical resection, with the option to go to surgery only if the tumor does not respond.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and complying with the protocol requirements and have signed the informed consent document. Patients with mild cognitive impairment may be considered for enrollment in the study if their legally authorized representative provides written informed consent for the patient.
* 18 years or older in age
* Biopsy proven dMMR (by IHC), Stage II or III colon cancer per CT imaging correlation with AJCC 8th edition, 2017, amendable to en block surgical resection as determined by colorectal surgeon.
* Biopsy specimen for diagnosis of dMMR Colon cancer should have enough tissue for minimum 4 and max 6 adjacent unstained FFPE slides (4µm each) as determined by Protocol Pathologist Dr. Anthony Snow for CD3+ and CD8+ analysis. If there is not enough tissue present in original sample, a repeat colonoscopy and biopsy may be performed; otherwise patient is not eligible.
* Potentially surgically resectable Stage II or III patients who are willing to forgo surgical resection if study endpoints are met. Patient with easily manageable bowel changes amenable to laxatives or stool softeners as outpatient per assessment by colorectal surgery are allowed. (See exclusion criteria #2)
* ECOG performance status less than or equal to 1
* Absence of metastatic disease on CT CAP with Contrast within 28 days from treatment start
* Absolute neutrophil count greater than or equal to 1,500/µL
* Platelets greater than or equal to 100,000/µL
* Hemoglobin greater than or equal to 9 g/dL
* Serum creatinine less than or equal to 1.5 x upper limit of normal (ULN) or calculated creatinine clearance 60mL/min using the Cockcroft-Gault equation
* Total bilirubin less than or equal to 1.5 x ULN (less than or equal to 2.0 in patients with known Gilberts syndrome) OR direct bilirubin less than or equal to 1 x ULN
* Aspartate aminotransferase and alanine aminotransferase less than or equal to 3.0 x ULN
* International normalized ratio (INR) or prothrombin time (PT) less than or equal to 1.5× ULN unless patient is receiving anticoagulant therapy if PT or partial thromboplastin (PTT) is within therapeutic range of intended use of anticoagulants. Activated partial thromboplastin time (aPTT) less than or equal to 1.5× ULN unless patient is receiving anticoagulant therapy if PT or PTT is within therapeutic range of intended use of anticoagulants
* Participants of childbearing potential must have a negative serum pregnancy test within 72 hours prior to taking study treatment and agree to use an adequate method of contraception from screening through 180 days after the last dose of study treatment. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner starting with first dose of study treatment through 180 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.

Exclusion Criteria:

* Synchronous primary tumor (i.e. more than 1)
* Obstruction or perforation requiring diverting ostomy or immediate resection, or bright red blood per rectum requiring urgent blood transfusion, from their primary tumor.
* Clinical T4b tumors
* Known hypersensitivity to dostarlimab components or excipients.
* Major surgery less than or equal to 3 weeks prior to initiating protocol therapy
* Received investigational therapy less than or equal to 3 months, or within a time interval less than at least 5 half- lives of the investigational agent, whichever is shorter, prior initiating protocol therapy.
* Heavy bleeding from the colon cancer tumors requiring PRBC transfusions that would require palliative surgical resection
* Concurrent, clinically significant, active malignancies within two years of study enrollment.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, glucocorticoids, or immunosuppressive drugs). Other than Replacement hormone therapy with thyroxine for hypothyroidism , insulin for T1 diabetes mellitus , or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.)
* Diagnosis of immunodeficiency or has received any systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days prior to initiating protocol therapy.
* History of greater than or equal to Grade 3 immune-related AE with prior immunotherapy, except for non-clinically significant lab abnormalities.
* Patients with known HIV (Human Immunodeficiency Virus) infection on effective retroviral therapy regardless of CD4 count who have had an opportunistic infection within the past 12 months.
* Organ transplant recipients on immunosuppressive medications
* Patients with chronic HBV infection with active disease who meet the criteria for anti HBV therapy but not on suppressive antiviral therapy prior to initiation of treatment of this protocol are excluded. Also, patients with history of HCV infection that have not completed curative antiviral treatment and the HCV viral load is not below the limit of quantification areexcluded.(e.g. a patient who is HCV Ab positive but HCV RNA negative due to prior treatment or natural resolution is eligible.)
* Prior history of interstitial lung disease.
* Received a live vaccine within 30 days of initiating protocol therapy.
* Not enough tissue for confirming dMMR status and CD3+ /CD8+ testing
* 19. Patients with severe cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Major Clinical Response (MCR) Rate | From Dostarlimab initiation to 18 weeks.
  MCR rate is defined as the proportion of patients meeting the following criteria at 18 weeks: 1) ctDNA is stable or declining, 2) a clinically asymptomatic primary tumor, and 3) no metastatic disease.

SECONDARY OUTCOMES:
Metastasis-Free Survival (MFS) Prior to Surgery | From Dostarlimab initiation until surgery or Dostarlimab completion, up to 2 years.
  MFS is defined as the time from treatment initiation to the date of metastasis or death due to any cause, if occurring prior to surgery. Otherwise, patients will be censored at the date of surgery or last radiographic assessment, whichever occurs first.
Progression-Free Survival (PFS) | From treatment Dostarlimab until study completion, up to 5 years.
  PFS is defined as the time from treatment initiation to the date of first documentation of disease progression (defined as increasing ctDNA, symptomatic primary tumor or metastasis), or death due to any cause. Otherwise, patients will be censored at last radiographic assessment.
Overall Response Rate (ORR) | From Dostarlimab initiation until surgery or Dostarlimab completion, up to 2 years.
  ORR is defined as the proportion of patients with RECIST disease response (CR, PR). All patients that do not meet the criteria for an objective response by the analysis cutoff date will be considered non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Saima M Sharif, MD, MS, Principal Investigator — University of Iowa Holden Comprehensive Cancer Center
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No